CLINICAL TRIAL: NCT03876418
Title: Surveillance, Prevention and Treatment of Intra-abdominal Hypertension and Abdominal Compartment Syndrome: A Single Center Prospective Cohort Study
Brief Title: Surveillance, Prevention and Treatment of Intra-abdominal Hypertension and Abdominal Compartment Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 100281
Record Dates: First submitted 2019-01-17; First posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Intra-Abdominal Hypertension; Abdominal Compartment Syndrome
MeSH Terms: conditions — Intra-Abdominal Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Patients undergo twice daily measurement of intra-abdominal pressure. Clinicians manage patients according to usual care.
- Aggressive (Active Comparator): Patients undergo aggressive surveillance (q6h) if intra-abdominal pressure is elevated as well as prevention and treatment according to protocol driven guidelines adapted from the World Society of the Abdominal Compartment. This may include nasogastric decompression, limiting fluid administration, drainage of ascites, paralysis and/or abdominal decompression.
  Interventions: Diagnostic Test: Intra-abdominal Pressure

INTERVENTIONS:
Diagnostic Test: Intra-abdominal Pressure — Aggressive screening, prevention and treatment of intra-abdominal hypertension
  Arms: Aggressive

SUMMARY:
This study evaluates the efficacy of intensive surveillance, prevention and treatment of intra-abdominal hypertension in ICU patients. In the first two months patients will be screened and undergo usual care. In the following 10-months patients will have more intensive screening and active measures towards prevention and treatment according to best practices.

DETAILED DESCRIPTION:
Elevated intra-abdominal pressures or intra-abdominal hypertension (IAH) has been shown to be common in all intensive care unit (ICU) patients (upwards of 50%) and has been suggested as the missing link in multi-organ dysfunction, and subsequently ICU mortality. Despite guidelines advocating prevention and surveillance of IAH, adherence remains low in most ICUs across North America and Europe.

The creation of the World Society of the Abdominal Compartment Syndrome (WSACS) in 2004 improved the recognition of IAH/ACS by intensivists. The first consensus guidelines from the WSACS were released in 2006, followed by a 2013 update. Additionally, clinical practice guidelines and recommendations for research were released in 2007 and 2009 respectively, which attempted to standardize research methods and reporting. Unfortunately, even in the 2013 guidelines only WEAK recommendations (by GRADE methodology) could be made regarding the efficacy of surveillance and treatment of IAH/ACS, citing a lack of high quality interventional trials.

The investigator's study aims to assess the feasibility of a larger multi-center interventional trial to investigate the efficacy of aggressive screening, prevention and treatment of IAH in ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 years of age)
* Admitted to intensive care unit
* Bladder catheter in-situ

Exclusion Criteria:

* Death prior to first IAP pressure measurement
* Pregnancy
* Expected ICU discharge within 24 hours
* Organ donor
* Clinical care team or patient/substitute decision maker declines to enroll patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days
  ICU Mortality

SECONDARY OUTCOMES:
% of bladder pressure measurements (feasibility) | 30 days
  Number of eligible measurements recorded / Number of eligible measurements
Length of stay | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Ian Ball, MD, Principal Investigator — London Health Sciences Center